CLINICAL TRIAL: NCT03692429
Title: An Open-label, Phase I Study to Assess the Safety of Multiple Doses of CYAD-101, Administered After Standard FOLFOX or FOLFIRI Chemotherapy in Patients With Unresectable Metastatic Colorectal Cancer
Brief Title: alloSHRINK - Standard cHemotherapy Regimen and Immunotherapy With Allogeneic NKG2D-based CYAD-101 Chimeric Antigen Receptor T-cells
Acronym: alloSHRINK
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-N2L-101
Record Dates: First submitted 2018-08-31; First posted 2018-10-02 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Unresectable Metastatic Colorectal Cancer
MeSH Terms: interventions — Folfox protocol; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYAD-101 with FOLFOX (Experimental): Infusion after standard FOLFOX chemotherapy
  Interventions: Drug: CYAD-101; Drug: FOLFOX
- CYAD-101 with FOLFIRI (Experimental): Infusion after standard FOLFIRI chemotherapy
  Interventions: Drug: CYAD-101; Drug: FOLFIRI

INTERVENTIONS:
Drug: CYAD-101 — Allogeneic NKG2D-based CYAD-101 Chimeric antigen Receptor T-cells
Drug: FOLFOX — 5-FU, leucovorin and oxaliplatin
  Arms: CYAD-101 with FOLFOX
Drug: FOLFIRI — 5-FU, leucovorin and irinotecan
  Arms: CYAD-101 with FOLFIRI

SUMMARY:
The purpose of the alloSHRINK study is to assess the safety, cell kinetics and clinical activity of CYAD-101 in patients with unresectable metastatic colorectal cancer administered after standard chemotherapy

DETAILED DESCRIPTION:
This Study aims to determine and confirm the recommended dose of the allogeneic CYAD-101 cells after standard FOLFOX or FOLFIRI chemotherapy in patients with unresectable metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven metastatic adenocarcinoma of the colon or rectum.

   1. Confirmed metastatic unresectable adenocarcinoma of the colon or the rectum.
   2. Recurrent/progressing disease after at least one line of systemic therapy for metastatic disease.
   3. Unequivocal and measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
   4. FOLFOX segment: Neurotoxicity less than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 from previous chemotherapy.
   5. FOLFIRI segment: Documented progressive disease (PD) under FOLFIRI treatment, with or without targeted therapy, given within 3 months prior to study registration. Anti-cancer therapy post FOLFIRI-documented PD prior to study registration is authorized if discontinued at least 7 days before the planned study registration. Radiotherapy is not authorized.
2. The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
3. The patient must have adequate bone marrow reserve, hepatic, renal, pulmonary and cardiac functions.

Exclusion Criteria:

1. The patient has a confirmed or history of tumor involvement in the central nervous system (CNS).
2. Any non-cancer-directed investigational agent within 3 weeks before the planned day for the first CYAD-101 administration.
3. Filgrastim (Granulocyte-Colony-Stimulating Factor [G-CSF]) or similar growth factors within 7 days before the planned day for the first CYAD-101 administration.
4. Prior allogeneic stem cell transplantation, chimeric antigen receptor therapy or other genetically modified T-cell therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-11-28 (Estimated); Study Completion 2036-02-17 (Estimated)

PRIMARY OUTCOMES:
Occurence of Dose Limiting Toxicities | Up to 82 days post first CYAD-101 Infusion

CONTACTS AND LOCATIONS:
Locations (4):
- Moffit Cancer Center, Tampa, Florida, United States
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michaux A, Mauen S, Breman E, Dheur MS, Twyffels L, Saerens L, Jacques-Hespel C, Gauthy E, Agaugue S, Gilham DE, Sotiropoulou PA. Clinical Grade Manufacture of CYAD-101, a NKG2D-based, First in Class, Non-Gene-edited Allogeneic CAR T-Cell Therapy. J Immunother. 2022 Apr 1;45(3):150-161. doi: 10.1097/CJI.0000000000000413. PMID 35191428